CLINICAL TRIAL: NCT05055115
Title: Ph.D.-Project: Eustachian Tube Dysfunction: Causes, Diagnosis, Treatment, and Prognosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Regional Hospital West Jutland (Other)
Responsible Party: Principal Investigator, Niels Højvang Holm, Principal Investigator. Doctor of Medicine. Ph.D.-student, Regional Hospital West Jutland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Niels Holm
Record Dates: First submitted 2021-08-31; First posted 2021-09-24 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Eustachian Tube Dysfunction; Middle Ear Disease; Hearing Loss, Conductive; Middle Ear Problem
Keywords: Balloon Eustachian Tuboplasty; Cone-beam computed tomography; CBCT; Eustachian Tube Dysfunction Questionnaire; ETDQ-7; Tubomanometry
MeSH Terms: conditions — Hearing Loss, Conductive

STUDY DESIGN:
Intervention Model Description: 50 patients will fill out the ETDQ-7 questionnaire before and after tympanostomy. Results will be compared to 50 age- and gender matched controls with no history of ETD or ear-surgery.
  Both MRI and Cone Beam-CT scans are performed in order to obtain a complete overview of ET. Twelve patients with ETD and 12 healthy controls are examined with both MRI and CBCT. The dimensions and angulations of the ET in the two groups are compared to identify significant differences.
  Tubomanometry is a tool to measures the dynamic function of the eustachian tube. 50 patients are examinated and compared to 50 controls to investigate tubomanometry's ability to distinguish the two groups.
  A REDCap-database is established in order to create a national cohort where all patients undergoing first time Balloon Eustachian Tuboplasty in Denmark, are registered. All patients are followed for 12 months. The patients, who benefit from the procedure, will be compared to those without effect.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Balloon Eustachian Tuboplasty (Experimental): Patients with long-lasting symptoms of ETD, who benefits from tympanostomy tube insertion, will be offered Balloon Eustachian Tuboplasty (BET) of the cartilaginous part of ET. The procedure is performed endonasally under general anesthesia. It is believed that BET leads to micro-bleeding in the mucosa with subsequent scarring and expansion of ET.
  Interventions: Procedure: Balloon Eustachian Tuboplasty

INTERVENTIONS:
Procedure: Balloon Eustachian Tuboplasty — Balloon Eustachian Tuboplasty of the cartilaginous part of ET. The procedure is performed endonasally under general anesthesia. It is believed that BET leads to micro-bleeding in the mucosa with subsequent scarring and expansion of ET.

SUMMARY:
Background:

The Eustachian Tube (ET) is a mucosa-lined connection between the nasopharynx and the middle ear cavity. It is believed to have three functions: 1) ventilation of and pressure equalization in the middle ear cavity, 2) mucus drainage from the middle ear, and 3) protection against sound and infection from the nasopharynx1. In adults, Eustachian Tube Dysfunction (ETD) can cause complaints from one or both ears. For many years, various definitions of ETD have been used, impairing the opportunity to compare studies. However, in 2015, an international consensus on definition, types, clinical presentation, and diagnosis of ETD was published by Schilder et al2, which has been adopted by all the Scandinavian countries. The symptoms include pressure (fullness), and/or pain in the ear, muffled hearing, and overall discomfort. Furthermore, chronic ETD can result in tympanic membrane retraction, atelectasis of the middle ear cavity, and ultimately formation of cholesteatoma3. Unfortunately, the symptoms of ETD are multiple and inaccurate giving rise to varying estimates of the prevalence. As an example, a study in UK found a 0.9 % prevalence of ETD4. In addition, clear guidelines on diagnostics and treatment are not currently available due to the fact, that no objective test for detection of ETD exists. In the need of a symptom scoring system, the patient reported Eustachian Tube Dysfunction Questionnaire (ETDQ-7) has been developed and validated in English5. Yet, translation into other languages as well as validation in other settings are necessary in order to substantiate the applicability of ETDQ-7. ETD is associated with a lack of opening of ET. It is believed that the length, diameter and angle of ET influences its ability to open regularly, thus affecting its function. A short, narrow and angled ET may predispose to ETD. However, the imaging available to visualize ET are not accurate enough to diagnose ETD. A direct test of the function of ET is not available. Tubomanometry is a relatively new method developed to directly test the opening of ET, but is yet to be validated6.

Both non-surgical and surgical treatment options to improve the function of the Eustachian Tube are available. Non-surgical management includes pressure equalization methods (e.g. the Valsalva maneuver), antihistamines, treatment with decongestants, and nasal douching with a saline solution. Surgically, ventilation tubes are often used to treat ETD. In case of adenoid hypertrophy obstructing the pharyngeal opening of ET, adenoidectomy is recommended. Balloon Eustachian Tuboplasty (BET) was introduced in 2010 by Ockermann et al7. BET is a non-invasive procedure performed under general anesthesia. During the procedure, a catheter is inserted either endonasally or transtympanic into ET, and a balloon is inflated with water for approximately two minutes. Various heterogeneous studies have shown a short-term effect of BET, but long-term effects are unclear8.

In summary, despite the assumption of being a common condition, the field of ETD suffers from lack of precise definition, diagnostic criteria, identification of underlying causes as well as purposeful treatment, and prognostic factors. Especially, long-term effects of BET need further investigation. Therefore, in an effort to fill out the gap of knowledge about ETD, the following specific aims are proposed:

DETAILED DESCRIPTION:
Specific Aims:

Translation, modification, and validation of the ETDQ-7 in Danish settings Investigation of combined Cone-Beam CT and MRI of the Eustachian tube in order to determine a potential anatomical cause/disposition of ETD Clarification of the effects of BET using strict criteria for ETD To validate the process of tubomanometry as an objective tool in patients with ETD

Hypothesis

ETDQ-7 is a useful patient-reported symptom scoring tool in Danish patients with assumed ETD ETD is related to the dimensions and angles of the Eustachian tube detected by combining Cone-Beat CT and MRI-scans BET is effective in patients with chronic ETD Tubomanometry can be used as an objective tool in diagnosing and monitoring the effect of treatment in patients with ETD.

Study 1:

Danish translation, modification, and validation of the Eustachian Tube Dysfunction Questionnaire Holm NH1 & Ovesen T1.

1) ENT Department, Regional Hospital West Jutland, Expected publication in Clinical Otolaryngology

The Eustachian Tube Dysfunction Questionnaire (ETDQ-7) was introduced in 2012 by McCloud et al. It scores symptoms of ETD, and it is the only validated patient-reported scoring tool. So far, ETDQ-7 has been translated and validated into German, Turkish, and Brazilian Portuguese. The aim of the present study is to translate, modify and validate the questionnaire in Danish settings to achieve a solid tool for optimal diagnostic and evaluation of treatment among patients with ETD.

Back and forth translation from English to Danish will be performed by a professional translator. Then, a modification/cultural adaption of the questionnaire will be conducted. Seventy-five patients older than 18 years referred to practicing ear nose and throat specialists will be included. Inclusion criteria are symptoms of ETD for more than three months including tympanometry compatible with negative middle ear pressure (C2 or B-curve). The seven questions in the ETDQ-7 are: 1) pressure in the ears, 2) pain in the ears, 3) a feeling that the ears are clogged or "under water", 4) ear symptoms when having a cold or sinusitis, 5) crackling or popping sound in the ears, 6) ringing in the ears or 7) feeling that the hearing is muffled. Patients will fill out the questionnaire before and after tympanostomy (insertion of ventilation tubes). Patients will then be referred to the ENT Department, Regional Hospital West Jutland for further follow up, including controlling the tympanostomy tubes. Here, a complete oto-rhino-laryngological examination, fiber optic naso-pharyngo-laryngo-scopy, pure tone audiometry, and tympanometry will be performed. SNOT-22 questionnaire is completed for differential diagnostics. Results will be compared to 75 age- and gender matched controls with no history of ETD or ear-surgery. In addition, patients undergoing BET will complete the questionnaire before and after surgery.

For test-retest data, 15 patients and 15 controls repeat filling out the questionnaire 14 days after the first reply. Patients are excluded from the retest in case of upper airway infection or travelling by airplane between the two tests. By comparing these results and calculating the Spearman's rank correlation coefficient, the test-retest reliability of ETDQ-7 is assessed. The internal consistency of the questionnaire will be investigated by using Cronbach's alpha coefficient and Spearman rho. Hence, it will be possible to conclude if ETDQ-7 can be used as a diagnostic tool to differentiate patients with ETD from individuals without ETD as well as to evaluate the effect of BET.

Study 2:

Cone-Beam CT combined with MRI as a diagnostic tool in patients with Eustachian Tube Dysfunction Holm NH1, Ovesen T1, Balazs M2 & Pedersen M3

1. ENT Department, Regional Hospital West Jutland
2. Department of Radiology, Regional Hospital West Jutland
3. Institute of Experimental Clinical Research, Aarhus University Hospital Expected publication in Otology and Neurotology

The Eustachian tube (ET) is both skeletal and cartilaginous in nature. CT and/or MRI are often used preoperatively to identify potential pathology in the temporal bone. However, these techniques are not routinely used in order to diagnose ETD. It is unclear whether ETD is associated pathology in the skeletal or cartilaginous regions of ET. Length, diameter and/or angle of the ET may be a potential anatomical explanation for ETD, alternatively a disposition of ETD.

Cone-beam computed tomography (CBCT) is a relatively new imaging technique, where divergent X-rays form a cone. CBCT can accurately visualize the facial bones, and is often used by dentists and orthodontics. A study has shown no difference in the temporal bone between patients with patulous Eustachian tube and a control group. No other study has investigated ETD patients with CBCT. The cartilaginous part of ET is ideally visualized with MRI, whereas CBCT is the best choice for the skeletal part. Both MRI and CBCT are therefore needed in order to obtain a complete overview of ET. By implementing a brand-new software technique, MRI and CBCT sequences will be fused. This will enable a better visualization of the ET, where the length, diameter and angle of ET can be measured more accurately than with the current available methods. Thus, dimensions of the ET in ETD patients can be classified accordingly to normal dimensions of ET.

To achieve this, twelve patients with ETD and 12 healthy controls are examined with both MRI and CBCT. The sequences will be fused and two radiologists will describe the scans blinded and independently. The dimensions and angulations of the ET in the two groups are compared to identify significant differences.

Study 3:

Balloon Eustachian Tuboplasty: indications and effect of treatment Holm NH1, Ovesen T1 & Sinkkonen ST2) 1) ENT Department, Regional Hospital West Jutland 2) Department of Otorhinolaryngology, Head and Neck Center, Helsinki University Hospital, Finland Expected publication in The Journal of Laryngology & Otology

Patients with long-lasting symptoms of ETD, who benefits from tympanostomy tube insertion, will be offered Balloon Eustachian Tuboplasty (BET) of the cartilaginous part of ET. The procedure is performed endonasally under general anesthesia. It is believed that BET leads to micro-bleeding in the mucosa with subsequent scarring and expansion of ET. Apparently, the procedure has a high success rate and low complication rate. Currently, little evidence exists regarding the long-term effects of BET, and it remains unclear which patients will benefit from the procedure.

The aim of this study is to create a national cohort where all patients undergoing first time BET in Denmark, are registered. A REDCap-database is established. All patients are followed for 12 months by ETDQ-7, oto-microscopy and tympanometry. The patients, who benefit from the procedure, will be compared to those without effect. Hence, the investigators hypothesize that it will be possible to assess which factors increase the probability of effect from BET in order to select patients for BET more accurately in the future.

Study 4:

Tubomanometry: an objective tool in diagnosing patients with Eustachian Tube Dysfunction Holm NH1, Ovesen T1 & Sudhoff H2

1) ENT Department, Regional Hospital West Jutland. 2) Klinikum Bielefeld, Head and Neck Surgery

Tubomanometry (TMM) was introduced in 2009 as an objective tool to measure the dynamic function of ET. While swallowing a small amount of water, a standardized air-pressure is applied through a nasal catheter. If the ET opens, pressure will be transferred to the middle ear cavity and the increased pressure will be measured with a probe in the ear channel. The test is harmless, relatively fast, and can be used even in case of perforation of the tympanic membrane or tympanostomy tube. In a control group, Schröder et al found an opening of ET in 97 %, opposed to 57 % in a group of ETD-patients. Another study showed that TMM has a high sensitivity, but low specificity for detecting ET opening. A reduced opening/lack of opening of ET is associated with ETD. Schilder et al concluded, that the existing evidence is weak, which is partly because of the disparate definitions of ETD. Finally, there is now consensus both internationally and in Denmark on definitions of ETD. Therefore, the investigators hope to develop new knowledge in an effort to develop a globally acceptable definition of ETD.

The investigators aim at examining 50 patients with ETD and compare them to 50 age- and gender matched controls to investigate TMM's ability to distinguish the two groups. The investigators believe that TMM has a great potential and most likely relates to the pathological process of the disease. It may be a useful tool in direct testing of the ET and monitoring the effect of treatment of ETD.

ELIGIBILITY:
Inclusion Criteria:

Patients are included in the study if they have presented constant or intermittent ETD symptoms for more than three months:

1. pressure in the ears,
2. pain in the ears,
3. a feeling that the ears are clogged or "under water",
4. ear symptoms when having a cold or sinusitis,
5. crackling or popping sound in the ears,
6. ringing in the ears,
7. feeling that the hearing is muffled.

Furthermore, objective signs of negative middle ear pressure are needed:

1. poorly retractable eardrum,
2. tympanometry compatible with negative middle ear pressure (C2 or B-curve).

Exclusion Criteria:

* patient refusal to participate in the study,
* head and neck surgery in the previous three months,
* head and neck irradiation,
* ETD symptoms <3 months,
* adenoid hypertrophy,
* nasal polyposis,
* acute upper respiratory infection or acute sinusitis,
* tympanic membrane perforation,
* age <18 years, cleft palate,
* craniofacial syndromes including Down's Syndrome,
* cystic fibrosis,
* ciliary dysmotility syndrome.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
ETDQ-7 | Up to12 months
  ETDQ-7 score before and after tympanostomy. ETDQ-7-score varies from 7 to 49 (higher score = worse symptoms)
Measurement of the eustachian tube | Up to 12 months
  The dimension (measured in mm) and the angle (degrees) of the Eustachian tube i measured by fusing ConeBeam CT and MRI-scans. The dimensions are then compared between groups of patients and controls.
Balloon Eustachian Tuboplasty | 12 months
  All patients undergoing BET are registered in a database and followed for 12 months by ETDQ-7, oto-microscopy and tympanometry. The patients, who benefit from the procedure, will be compared to those without effect. Hence, the investigators hypothesize that it will be possible to assess which factors increase the probability of effect from BET in order to select patients for BET more accurately in the future.
  The ETDQ-7-score varies from 7 to 49 (higher score = worse symptoms)
R-value measured with tubomanometry in patients and controls | Up to 12 months
  Tubomanometry examines the opening of the Eustachian tube and is measured with a R-score, ranging from 0 to infinite. The R-score is grouped into three: a normal opening (R<1), delayed opening (R>1) and no opening R = 0. If the opening is delayed or doesn't happen, it indicates an dysfunction of the Eustachian tube. The investigators aim at examining 50 patients with ETD and compare them to 50 age- and gender matched controls to investigate the ability of tubomanometry to distinguish the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Niels H. Holm, MD, Principal Investigator — Hospitalsenheden Vest
Locations (1):
- Regional Hospital West Jutland, Holstebro, Denmark

REFERENCES:
- [Derived] Holm NH, Ovesen T. The Usefulness of ETDQ-7 Score in Assessing ETD. Clin Otolaryngol. 2025 Sep;50(5):840-847. doi: 10.1111/coa.14324. Epub 2025 Apr 25. PMID 40276950